CLINICAL TRIAL: NCT01643187
Title: Comparison of the Effect of Two Treatments on the Nutritional and Micronutrient Status of Malnourished Children From the Takalik Abaj
Brief Title: Comparison of the Effect of Two Treatments on the Nutritional and Micronutrient Status of Malnourished Children
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Association for the Study and Prevention of HIV/AIDS (Other)
Responsible Party: Principal Investigator, Victor Alfonso Mayen, Nutritionist, Magister Science, Association for the Study and Prevention of HIV/AIDS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APE-001
Record Dates: First submitted 2012-07-13; First posted 2012-07-18 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Minerals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fortified beverage (Experimental): A group of children with some degree of malnourishment considered by a Z-score < -1 for weight for height, height for age or weight for age.
  Interventions: Dietary Supplement: Beverage fortified with 21 vitamins and minerals
- Group receiving lactose-free milk (Active Comparator): A group of children with some degree of malnourishment considered by a Z-score < -1 for weight for height, height for age or weight for age.
  Interventions: Dietary Supplement: Lactose-free milk

INTERVENTIONS:
Dietary Supplement: Beverage fortified with 21 vitamins and minerals — The serving contains 4 grs. of protein, 12 grs. of carbohydrate, 1 gr of fat 9 mg of zinc, 12.5 mg iron, 160 µg of folic acid, 90 µg of iodine, 250 mg of vitamin A, 40 mg of vitamin C, 0.5 mg of vitamin B6, 0.9 µg of vitamin B12, 6 mg of niacin, 0.5 mg of vitamin B2, 0.5 mg of vitamin B1, 0.3 mg of copper, 5 mg of vitamin D3, 5 mg of vitamin E, 200 mg ofcalcium, 150 mg of phosphorous, 40 mg of magnesium, 17 µg of selenium, 0.17 µg of manganese, 1.8 mg of pantothenic acid and 8 µg of biotin.
  Other Names: Chispuditos®
  Arms: Fortified beverage
Dietary Supplement: Lactose-free milk — Serving contains 4 grs. of protein, 12 grs of carbohydrate and 1 gr of fat
  Other Names: High nutritive value vegetable mix
  Arms: Group receiving lactose-free milk

SUMMARY:
The purpose of this study is to measure the impact of a fortified food on the nutritional and micronutrient status of malnourished children, compared with milk. The changes to be evaluated include the indicators weight for height, height for age, weight for age, mid-arm circumferance for age; and levels of hemoglobin, serum zinc, serum ferritin, serum folic acid, erythrocyte folic acid, serum vitamin B12, and urinary iodine.

DETAILED DESCRIPTION:
Chronic malnutrition evidenced by short height for age is a common nutritional problem in underdeveloped countries which is generally accompanied by iron deficiency anemia and zinc deficiency. It has many consequences on the adult including limited capacity to work and higher risk of obesity and chronic disease. The present study will offer a fortified food, culturally accepted and locally produced. The effectiveness of this fortified food compared to lactose-free milk, in a controlled dose and with no risk to the health of the study participants, will be determined. Both will be distributed for free to be consumed as an atole or in liquid form, respectively, at a community level in an environment controlled as much as possible. This will allow to determine adherence, acceptability, consumption and distribution within the family.

ELIGIBILITY:
Inclusion Criteria:

* Some degree of malnutrition according to weight for height or height for age
* Reside in one of the six communities chosen for the study

Exclusion Criteria:

* Leukemia
* Diabetes
* Handicap
* Down syndrome
* Renal failure

Ages: 6 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change in Nutritional status | Months 0, 3, 6, 9, 12 and 15 months
  weight for height Z-score, height for age Z-score, weight for age Z-score and mid arm circumferance

SECONDARY OUTCOMES:
Iron Status | Months 0 and 16
  Hemoglobin level and serum ferritin level
Zinc status | Months 0 and 16
  serum zinc level

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reinhart, Study Chair — Mathile Institute
Locations (1):
- APEVIHS, Retalhuleu, Guatemala

REFERENCES:
- [Result] Brown KH, Peerson JM, Rivera J, Allen LH. Effect of supplemental zinc on the growth and serum zinc concentrations of prepubertal children: a meta-analysis of randomized controlled trials. Am J Clin Nutr. 2002 Jun;75(6):1062-71. doi: 10.1093/ajcn/75.6.1062. PMID 12036814
- [Result] Ministry of Social Health and Public Assistance et al. Micronutrient National Survey. Guatemala MSPAS 56pp. 2011
- [Result] Ministry of Public Health and Social Assistance. Maternal Infant Health Survey. Guatemala, MSPAS, 634 pp. 2010